CLINICAL TRIAL: NCT04721223
Title: A Phase 1b/2a, Multi-Center, Open-Label，Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of JAB-3068 in Combination With JS001 in Patients With Advanced Solid Tumors
Brief Title: JAB-3068 Activity in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-3068-03
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumor; Esophageal Squamous Cell Carcinoma; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JAB-3068+PD1 inhibitor Part1 (Experimental): JAB-3068+JS001 dose escalation
  Interventions: Drug: JAB-3068; Drug: PD1 inhibitor
- JAB-3068+PD1 inhibitor Part2 (Experimental): JAB-3068+JS001 dose expansion
  Interventions: Drug: JAB-3068; Drug: PD1 inhibitor

INTERVENTIONS:
Drug: JAB-3068 — JAB-3068 administrated orally as a tablet.
Drug: PD1 inhibitor — JS001 administrated as an intravenous(IV) infusion.

SUMMARY:
To evaluate the safety and tolerability of JAB-3068 administered in investigational regimens in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
To assess the safety and tolerability and determine the recommended phase 2 dose (RP2D) of JAB-3068 in combination with PD1 inhibitor in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, according to local guidelines, signed and dated by the participant prior to the performance of any study-specific procedures, sampling, or analyses.
* Participant must be ≥18 years of age at the time of signature of the informed consent form (ICF).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

Exclusion Criteria:

* History (≤3 years) of cancer that is histologically distinct from the cancers under study, except for cervical carcinoma in situ, superficial non-invasive bladder tumors, or curatively treated Stage I non-melanoma skin cancer
* Known serious allergy to experimental drugs
* Brain or spinal metastases, except if treated by surgery, surgery plus radiotherapy or radiotherapy alone, with no evidence of progression or hemorrhage for ≤21 days before the start of treatment with the study drugs, and has not received any systemic corticosteroids for ≥21 days before the start of treatment with the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | 24 months
  Incidence of dose limiting toxicities (DLTs) . A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle with JAB-3068 and JS001.
Objective response rate (ORR) | 24 months
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR).

SECONDARY OUTCOMES:
Plasma concentration (Cmax) | 24 months
  Highest observed plasma concentration of JAB-3068 and JS001
Time to achieve Cmax (Tmax) | 24 months
  Time of highest observed plasma concentration of JAB-3068 and JS001
Area under the plasma concentration-time curve (AUC) | 24 months
  Area under the plasma concentration time curve of JAB-3068 and JS001
Duration of response ( DCR ) | 24 months
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD).
Progression-free survival (PFS) | 24 months
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first.
Duration of response ( DOR ) | 24 months
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | 24 months
  OS is defined as the interval of time between the date of first treatment until death, loss to follow up or termination of the study by the sponsor.
Number of Participants with Treatment-related Adverse Events(TRAE) | 24 months
  TRAE is defined as the AES that the casual relationship of the AE is ralated to investigational drug.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No